CLINICAL TRIAL: NCT01730482
Title: A Phase 1 Study to Investigate the Absorption, Metabolism and Excretion of [14C] AT1001 (Migalastat Hydrochloride) Following a Single Oral Administration in Healthy Volunteers (AT1001-014)
Brief Title: A Study to Assess the Absorption, Metabolism and Excretion of Migalastat Hydrochloride (AT1001-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116435
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Fabry Disease
Keywords: excretion; healthy volunteer; migalastat hydrochloride; AT1001; pharmacokinetics; Fabry disease
MeSH Terms: conditions — Fabry Disease | interventions — larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C] AT1001 Arm (Experimental): Each subject will receive a single oral dose of 150 mg of [14C] AT1001 as an aqueous solution containing 1 μCi AT1001 on Study Day 1.
  Interventions: Drug: [14C] AT1001

INTERVENTIONS:
Drug: [14C] AT1001 — 150 mg of [14C] labelled AT1001 will be administered as a solution (prepared by weighing 150 mg of AT1001 powder and dissolving in 100 mL of water). The entire solution will be swallowed orally. After ingestion of study medication, the dosing bottle will be rinsed with 50 mL of water and this will be ingested by the subject. This rinse procedure should be performed twice. Following the second rinse ingestion, the subjects should be instructed to drink additional water to bring the total volume ingested to 240 mL.

SUMMARY:
This study is designed to describe the metabolism of AT1001 (migalastat HCl) and the contribution of metabolism and urinary excretion to its overall elimination as part of the continuing assessment of the safety and effectiveness of the drug.

This is a Phase 1, single-site, open-label, single dose study of the absorption, metabolism and excretion of radiolabeled AT1001 in healthy male subjects between 30 and 55 years of age, inclusive. Six subjects will be dosed, with the goal of having at least 4 subjects complete the study through follow-up. All subjects will be screened within 28 days before admission to the Clinical Unit. Subjects will be confined to the clinical unit for 10 days after dosing and will return to the clinic for a follow-up visit 28 days after dosing.

Each subject will receive a single oral dose of AT1001 as an aqueous solution containing 150 mg [14C] AT1001 (1 μCi). Blood, duodenal bile, expired air, urine, and feces samples will be collected at specified time points after dosing throughout the period of confinement at the study site. Safety will be assessed throughout the study by monitoring clinical laboratory tests, ECGs, physical examinations, vital signs, and adverse events. The total duration of the study for each subject is approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 30 and 55 years, inclusive
* Body mass index (BMI) of >=18.0 to <=30.0 and weighing at least 60 kg
* Anticipated, regular, average bowel movements of 1-2 per day
* No clinically significant abnormal findings on the physical exam, vital signs, serum chemistry, hematology, and urinalysis values, as deemed by the principal investigator
* Willing to avoid taking of all over-the-counter medications 7 days and all prescription drugs 14 days prior to Day -1
* Willing to abstain from sexual intercourse or employ a barrier method of contraception during the inpatient clinic confinement and until the follow-up visit
* Willing to avoid ingestion of broccoli, brussels sprouts, grapefruit, grapefruit juice, or charbroiled meat during the period of confinement in the clinical unit
* Willingness to consume a fiber-rich diet during the period of confinement in the clinic
* Willingness to avoid vigorous physical activity during inpatient clinic confinement and through the follow-up visit
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, other study procedures, and study restrictions
* Provide written informed consent to participate in the study

Exclusion Criteria:

* Any previous or ongoing clinically significant illness, medical condition, medical history, physical findings, ECG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the subject, or alter the absorption, distribution, metabolism, or excretion of the study drug, or could impair the assessment of study results
* History or presence of significant ophthalmic, cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease
* History of a major surgical procedure within 30 days before screening
* History of blood or plasma donation or blood loss (>400 mL) within 60 days before screening
* History of drug or alcohol abuse or addiction within 2 years before screening
* Intake of more than 2 alcoholic drinks per day within the past 7 days or use of alcohol-, grapefruit-, or caffeine-containing foods or beverages within 72 hours prior to Day -1
* Self-reported smoker (occasional or frequent) or positive urine cotinine test (measured at screening and baseline) exceeding the local laboratory's lower limit of detection.
* Presence or history of severe adverse reaction to any drug; history of hypersensitivity or allergic reaction to AT1001 or related iminosugars
* Receipt of any investigational agent or participation in any other interventional clinical trial within the past 30 days
* Participation in any clinical study involving administration of [14C] labeled compound(s) within the last 12 months. A subject's previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study
* At Day -1, a drug toxicology screen positive for any illicit substances, or alcohol
* Anticipated need for alcohol, tobacco, or any drug during the period of confinement in the clinical unit

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Recovery of total radioactivity in urine | Days 1 to 11
  Urine will be collected: pre-dose (-12-0 hours), 0-12 and 12-24 hours on Day 1, 24-hourly on Days 2-10; the last sample will be collected on Day 11. Total radioactivity excreted in urine will be calculated for the entire collection period. The excretion rate will be calculated from total radioactivity collected in urine, divided by the duration of collection. The percentage of dose excreted in urine will be calculated from the total amount excreted in urine divided by the dose administered, multiplied by 100.
Recovery of total radioactivity in feces | Days 1 to 11
  Feces will be collected: predose (-24 to 0 hours); all bowel movements post-dose will be collected on Days 1 to 10; the last sample will be collected on Day 11. Total radioactivity excreted in feces will be calculated for the entire collection period. The excretion rate will be calculated from total radioactivity collected in feces, divided by the duration of collection. The percentage of dose excreted in feces will be calculated from the total amount excreted in feces divided by the dose administered, multiplied by 100.
Presence of radioactivity in expired air | Day 1
  Expired air will be collected: pre-dose and at 2, 4, 6 and 24 hours after dosing. Each subject will blow into a measured volume of sodium hydroxide solution containing phenolphthalein, until an indicator changes color, showing that the sodium hydroxide is saturated. This sodium hydroxide solution will be analysed for radioactive content. If radioactivity is detected the total amount in expired air during the collection period will be calculated.
Plasma AT1001 pharmacokinetic parameters | Days 1 to 10
  Blood samples will be collected: Pre-dose, at 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 and 240 hours after dosing. Non-compartmental pharmacokinetic parameters will be calculated for plasma AT1001: area under the drug concentration-time curve (AUC) from time zero to the time of the last measurable concentration, AUC from time zero to infinity, maximum observed drug concentration, time of the maximum drug concentration, apparent terminal elimination rate constant and apparent elimination half life.
Plasma total radioactivity pharmacokinetic parameters | Days 1 to 10
  Blood samples will be collected: Pre-dose, at 30 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 and 240 hours after dosing. Non-compartmental pharmacokinetic parameters will be calculated for plasma radioactivity: area under the drug concentration-time curve (AUC) from time zero to the time of the last measurable concentration, AUC from time zero to infinity, maximum observed drug concentration, time of the maximum drug concentration, apparent terminal elimination rate constant and apparent elimination half life.

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Day 1 to Day 29
  Adverse events (AEs) will be collected from the start of Investigation Product and until the follow-up visit.
Measure of clinical laboratory test values to access safety and tolerability | Upto 8 weeks
  Clinical laboratory tests will include hematology, coagulation tests, clinical chemistry, urinalysis, drug and toxicology screen, Hepatitis A and HIV screen.
Physical examination to access safety and tolerability | Upto 8 weeks
  Physical examination results will be categorized as normal, abnormal clinically significant, or abnormal not clinically significant
Measure of vital signs to access safety and tolerability | Upto 8 weeks
  Vital sign measurements will include pulse, respiratory rate, blood pressure, and oral temperature). Subjects should be in a supine position for at least 5 minutes prior to taking measurements.
Measure of ECG to access safety and tolerability | Upto 8 weeks
  Electrocardiograph (ECG) is a machine that measures the electrical activity of the heart and records changes in the hearts' rhythm. All subjects will undergo ECG testing.
The blood to plasma ratio of total radioactivity | Day 1
  The ratio of plasma to blood radioactivity will be calculated at 2, 4, 6 and 24 hours after administration of AT1001.
Characterization of metabolites in plasma, urine, duodenal bile and fecal homogenates | Day -1 to Day 11
  An Entero-Test capsule will be ingested to collect duodenal bile and will be removed after sample collection. Metabolite elucidation and identification will be performed in the collected plasma, urine doudenal bile, and fecal samples, if feasible, under a separate study. Results will be summarized in a separate report.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics